CLINICAL TRIAL: NCT01176266
Title: An Open-Label, Multicenter, Multinational Study of the Safety, Efficacy and Pharmacokinetics of Asfotase Alfa (Human Recombinant Tissue-nonspecific Alkaline Phosphatase Fusion Protein) in Infants and Children ≤ 5 Years of Age With Hypophosphatasia (HPP)
Brief Title: Open-Label Study of Asfotase Alfa in Infants and Children ≤ 5 Years of Age With Hypophosphatasia (HPP)
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Alexion Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ENB-010-10
Record Dates: First submitted 2010-07-29; First posted 2010-08-05 (Estimated); Results first posted 2018-02-26 (Actual); Last update posted 2019-03-13 (Actual); Status verified 2019-03

CONDITIONS: Hypophosphatasia
Keywords: Hypophosphatasia; HPP; Bone Disease; Soft Bones; Low Alkaline Phosphatase; Genetic metabolic disorder; Alkaline phosphatase; Tissue-specific alkaline phosphatase (TNSALP); Rickets; Osteomalacia
MeSH Terms: conditions — Hypophosphatasia; Bone Diseases; Rickets; Osteomalacia | interventions — asfotase alfa

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Asfotase alfa (Experimental): A total of 6 mg/kg/week of asfotase alfa administered by SC injection (either 1 mg/kg asfotase alfa 6 times per week, or 2 mg/kg asfotase alfa 3 times per week)
  Interventions: Drug: asfotase alfa

INTERVENTIONS:
Drug: asfotase alfa
  Other Names: ENB-0040

SUMMARY:
This clinical trial was conducted to study hypophosphatasia (HPP), a bone disorder caused by gene mutations or changes. These gene mutations cause low levels of an enzyme needed to harden bone. The purpose of this study was to test the safety and efficacy of a study drug called asfotase alfa (human recombinant tissue non-specific alkaline phosphate fusion protein) to see what effects it has on patients 5 years of age or less with HPP.

DETAILED DESCRIPTION:
Asfotase alfa was formerly referred to as ENB-0040

Hypophosphatasia (HPP) is a life-threatening, genetic, and ultra-rare metabolic disease characterized by defective bone mineralization and impaired phosphate and calcium regulation that can lead to progressive damage to multiple vital organs, including destruction and deformity of bones, profound muscle weakness, seizures, impaired renal function, and respiratory failure. There are limited data available on the natural course of this disease over time, particularly in patients with the juvenile-onset form.

ELIGIBILITY:
Inclusion Criteria:

Patients must meet all of the following criteria for enrollment in this study:

1. Parent or legal guardian(s) must provide written informed consent prior to any study procedures being performed and must be willing to comply with all study-required procedures. Where appropriate and required by local regulations, patient assent should also be provided prior to any study procedures being performed.
2. Documented diagnosis of HPP as indicated by:

   1. Total serum alkaline phosphatase (ALP) below the lower limit of normal for age NOTE: Historical values for ALP may be used to determine patient eligibility.
   2. Plasma pyridoxal-5'-phosphate (PLP) above the upper limit of normal (unless patient is receiving pyridoxine for seizures) NOTE: Historical values for PLP may be used to determine patient eligibility.
   3. Radiographic evidence of HPP at screening, characterized by:

      * Flared and frayed metaphyses, and
      * Severe, generalized osteopenia, and
      * Widened growth plates, and
      * Areas of radiolucency or sclerosis
   4. Two or more of the following HPP-related findings:

      * History or presence of: i) Nontraumatic post-natal fracture or ii) Delayed fracture healing
      * Nephrocalcinosis or history of elevated serum calcium
      * Functional craniosynostosis
      * Respiratory compromise or rachitic chest deformity
      * Vitamin B6-responsive seizures
      * Failure to thrive
3. Onset of symptoms prior to 6 months of age
4. Chronological age or adjusted age for premature infants born ≤ 37 weeks gestation of ≤ 5 years
5. Otherwise medically stable in the opinion of the Investigator and/or Sponsor

Exclusion criteria:

Patients will be excluded from enrollment in this study if they meet any of the following exclusion criteria:

1. Clinically significant disease that precludes study participation, in the opinion of the Investigator and/or Sponsor
2. Serum calcium or phosphate levels below the normal range
3. Current evidence of treatable form of rickets
4. Prior treatment with bisphosphonates
5. Treatment with an investigational drug within 1 month prior to the start of asfotase alfa treatment
6. Current enrollment in any other study involving an investigational new drug, device or treatment for HPP (e.g., bone marrow transplantation)
7. Intolerance to the investigational product (IP) or any of its excipients
8. Previous participation in the same study
9. Family relative of the Investigator

Ages: 1 Minute to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 69 (Actual)
Dates: Start 2010-07; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (23):
- United States (3):
  - Children's Hospital & Research Center Oakland, Oakland, California
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania
- Australia (2):
  - Lady Cilento Children's Hospital, South Brisbane, Queensland
  - Royal Children'S Hospital Melbourne, Parkville, Victoria
- Health Sciences Centre Winnipeg, University of Manitoba, Winnipeg, Manitoba, Canada
- France (2):
  - Necker Hospital, Paris
  - Chu de Toulouse, Toulouse
- Universitätskinderklinikum Würzburg, Würzburg, Germany
- Italy (2):
  - Istituto Giannina Gaslini, Genova
  - Ospedale Pediatrico Bambino Gesù, Roma
- Japan (5):
  - Fukuoka Higashi Medical Hospital, Koga, Fukuoka
  - Ishikawa Prefectural Hospital, Kanazawa, Ishikawa-ken
  - St. Marianna University School of Medicine, Yokohayama City Seibu Hospital, Yokohama, Kanagawa
  - Tokyo Medical University Hospital, Shinjuku, Tokyo
  - Saitama Municipal Hospital, Saitama
- Federal State Budgetary Institution, Moscow, Russia
- King Faisal Specialist Hospital and Research Center, Riyadh, Saudi Arabia
- Hospital Infantil Universitario Nino Jesus, Madrid, Spain
- Uludag University, Bursa, Turkey (Türkiye)
- United Kingdom (3):
  - Birmingham Children's Hospital, Birmingham
  - Royal Manchester Children'S Hospital, Manchester
  - Sheffield Children'S Hospital, Sheffield

REFERENCES:
- [Derived] Padidela R, Yates R, Benscoter D, McPhail G, Chan E, Nichani J, Mughal MZ, Myer C 4th, Narayan O, Nissenbaum C, Wilkinson S, Zhou S, Saal HM. Characterization of tracheobronchomalacia in infants with hypophosphatasia. Orphanet J Rare Dis. 2020 Aug 6;15(1):204. doi: 10.1186/s13023-020-01483-9. PMID 32762706
- [Derived] Hofmann CE, Harmatz P, Vockley J, Hogler W, Nakayama H, Bishop N, Martos-Moreno GA, Moseley S, Fujita KP, Liese J, Rockman-Greenberg C; ENB-010-10 Study Group. Efficacy and Safety of Asfotase Alfa in Infants and Young Children With Hypophosphatasia: A Phase 2 Open-Label Study. J Clin Endocrinol Metab. 2019 Jul 1;104(7):2735-2747. doi: 10.1210/jc.2018-02335. PMID 30811537
- [Derived] Whyte MP, Rockman-Greenberg C, Ozono K, Riese R, Moseley S, Melian A, Thompson DD, Bishop N, Hofmann C. Asfotase Alfa Treatment Improves Survival for Perinatal and Infantile Hypophosphatasia. J Clin Endocrinol Metab. 2016 Jan;101(1):334-42. doi: 10.1210/jc.2015-3462. Epub 2015 Nov 3. PMID 26529632
- See also: HPP support group — http://www.magicfoundation.org
- See also: US Hypophosphatasia Group (Soft Bones) — http://www.softbones.org
- See also: Hypophosphatasia Website — http://www.hypophosphatasia.com
- See also: Hypophosphatasia Website for Healthcare Providers — http://www.hypophosphatasia.com/hcp/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The main criteria for inclusion in the study were male and female patients less than or equal to 5 years of age with a documented diagnosis of infantile onset hypophosphatasia (HPP) who were otherwise medically stable. Patients must have had onset of HPP signs/symptoms prior to 6 months of age.
Period: Overall Study
Arm/Group | Asfotase Alfa
Started | 69
Completed | 60
Not Completed | 9
Not completed — Death | 6
Not completed — Withdrawal by Subject | 3

BASELINE CHARACTERISTICS:
Population: Full Analysis Set (defined as all patients who received any asfotase alfa treatment)
Arm/Group | Asfotase Alfa
Number analyzed (Participants) | 69
Age, Continuous [Mean (Standard Deviation); unit: weeks] | 113.42 (108.912)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36
  Male | 33
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 63
  Unknown or Not Reported | 5
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaskan Native | 0
  Asian | 7
  Black or African American | 0
  Native Hawaiian or Other Pacific Islander | 0
  White | 54
  Other | 3
  Unknown | 5

OUTCOME MEASURES:

1. Primary Outcome: Effect of Asfotase Alfa Treatment on Skeletal Manifestations of Hypophosphatasia (HPP)
Description: The effect of asfotase alfa treatment on skeletal manifestations of HPP (i.e., change in rickets severity) was measured by radiographs using a qualitative Radiographic Global Impression of Change (RGI-C) scale. Skeletal radiographs obtained at Week 24 were compared with skeletal radiographs obtained before initiation of treatment. The RGI-C is a 7-point rating scale that ranges from -3 (indicative of severe worsening of HPP-associated rickets) to +3 (indicative of complete or near complete healing of HPP-associated rickets).
Time Frame: From Baseline to Week 24
Population: Full Analysis Set
Measure: Median (Full Range); unit: scores on a scale
Arm/Group | Asfotase Alfa
Number analyzed (Participants) | 69
scores on a scale | 2.00 [-1.67 to 3.00]

2. Primary Outcome: Safety and Tolerability of Repeated Subcutaneous (SC) Injections of Asfotase Alfa
Description: Safety and tolerability of repeated subcutaneous (SC) injections of asfotase alfa for all treated patients was assessed by the number of patients with 1 or more treatment-emergent adverse event.
Time Frame: Up to 72 months or until regulatory approval in the country of residence. Patients received study drug for a median duration of 829.0 days, with a range from 6 to 2116 days (ie, from 0.9 week to 5.8 years).
Population: Full Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | Asfotase Alfa
Number analyzed (Participants) | 69
Participants | 69

3. Secondary Outcome: Effect of Asfotase Alfa Treatment on Skeletal Manifestations of Hypophosphatasia (HPP)
Description: The effect of asfotase alfa treatment on skeletal manifestations of HPP (i.e., change in rickets severity) was measured by radiographs using a qualitative Radiographic Global Impression of Change (RGI-C) scale. Skeletal radiographs obtained at the patient's last assessment were compared with skeletal radiographs obtained before initiation of treatment. The RGI-C is a 7-point rating scale that ranges from -3 (indicative of severe worsening of HPP-associated rickets) to +3 (indicative of complete or near complete healing of HPP-associated rickets).
Time Frame: Up to 72 Months or regulatory approval in the country of residence. Patients received study drug for a median duration of 829.0 days, with a range from 6 to 2116 days (ie, from 0.9 week to 5.8 years).
Population: Full Analysis Set
Measure: Median (Full Range); unit: scores on a scale
Arm/Group | Asfotase Alfa
Number analyzed (Participants) | 67
scores on a scale | 2.33 [-2.67 to 3.00]

4. Secondary Outcome: Effect of Asfotase Alfa Treatment on Ventilator-free Survival (Week 312)
Description: For patients who were not on respiratory support at the time of enrollment, the Kaplan-Meier estimate of ventilator-free survival at the end of the study
Time Frame: as for outcome 2
Population: Patients on respiratory support at Baseline were excluded from the analysis.
Measure: Number; unit: Probability
Arm/Group | Asfotase Alfa
Number analyzed (Participants) | 45
Probability | 0.81

5. Secondary Outcome: Effect of Asfotase Alfa Treatment on Respiratory Function
Description: Effect of asfotase alfa treatment on respiratory function as measured by the shift in proportion of patients requiring respiratory support at their last assessment compared with Baseline.
Time Frame: as for outcome 2
Population: Full Analysis Set
Measure: Count of Participants; unit: Participants
Groups:
- Baseline: Baseline assessment before initiation of asfotase alfa
- Asfotase Alfa - Without Respiratory Support at Baseline: Results at End of Study for Those Without Respiratory Support at Baseline (Last Assessment for Each Patient)
- Asfotase Alfa - With Respiratory Support at Baseline: Results at End of Study for Those With Respiratory Support at Baseline (Last Assessment for Each Patient)
Arm/Group | Baseline | Asfotase Alfa - Without Respiratory Support at Baseline | Asfotase Alfa - With Respiratory Support at Baseline
Number analyzed (Participants) | 69 | 45 | 24
Participants
  No respiratory support | 45 | 43 | 11
  Supplemental oxygen | 6 | 1 | 2
  Biphasic positive airway pressure | 0 | 0 | 0
  Continuous positive airway pressure | 4 | 1 | 2
  Mechanical ventilation | 13 | 0 | 9
  Other | 1 | 0 | 0

6. Secondary Outcome: Effect of Asfotase Alfa Treatment on Physical Growth - Length/Height Z-scores Change From Baseline to Last Obtained Value
Description: Effect of asfotase alfa treatment on physical growth as measured by change from Baseline to last assessment for each patient in length/height Z-scores
Time Frame: as for outcome 2
Population: Full Analysis Set
Measure: Median (Full Range); unit: Z-score
Arm/Group | Asfotase Alfa
Number analyzed (Participants) | 66
Z-score | 0.5 [-4 to 4]

7. Secondary Outcome: Effect of Asfotase Alfa Treatment on Physical Growth - Weight Z-scores Change From Baseline to Last Obtained Value
Description: Effect of asfotase alfa treatment on physical growth as measured by change from Baseline to last assessment for each patient in weight Z-scores
Time Frame: as for outcome 2
Population: Full Analysis Set
Measure: Median (Full Range); unit: Z-score
Arm/Group | Asfotase Alfa
Number analyzed (Participants) | 67
Z-score | 1.0 [-5 to 6]

8. Secondary Outcome: Effect of Asfotase Alfa on Biomarkers - Plasma Inorganic Pyrophosphate (PPi) Change From Baseline to Last Obtained Value
Description: Effect of asfotase alfa on PPi as measured by change from Baseline to last assessment for each patient
Time Frame: as for outcome 2
Population: Full Analysis Set
Measure: Median (Full Range); unit: uM
Arm/Group | Asfotase Alfa
Number analyzed (Participants) | 63
uM | -2.460 [-12.18 to 22.47]

9. Secondary Outcome: Effect of Asfotase Alfa on Biomarkers - Plasma Pyridoxal-5' Phosphate (PLP) Change From Baseline to Last Obtained Value
Description: Effect of asfotase alfa on PLP as measured by change from Baseline to last assessment for each patient
Time Frame: as for outcome 2
Population: Full Analysis Set
Measure: Median (Full Range); unit: ng/mL
Arm/Group | Asfotase Alfa
Number analyzed (Participants) | 56
ng/mL | -395.40 [-23836.0 to 2400.0]

10. Secondary Outcome: Effect of Asfotase Alfa on Serum Parathyroid Hormone (PTH) - Change From Baseline to Last Obtained Value
Description: Effect of asfotase alfa on serum PTH as measured by change from Baseline to last assessment for each patient
Time Frame: as for outcome 2
Population: Full Analysis Set
Measure: Median (Full Range); unit: pmol/L
Arm/Group | Asfotase Alfa
Number analyzed (Participants) | 47
pmol/L | 0.70 [-4.7 to 5.7]

11. Secondary Outcome: Effect of Asfotase Alfa Treatment on Tooth Loss
Description: Effect of asfotase alfa treatment on tooth loss assessed by the proportion of patients who experienced tooth loss during the study
Time Frame: as for outcome 2
Population: Full Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | Asfotase Alfa
Number analyzed (Participants) | 69
Participants | 42

12. Secondary Outcome: Pharmacokinetic (PK) Properties of Asfotase Alfa (Tlast)
Description: The PK properties (tlast) of asfotase alfa
Time Frame: PK parameters were calculated using Week 6 study visit data. Week 6 study visit blood samples for PK testing were drawn pre-dose and 6, 12, 24, 32, and 48 hours post dose
Population: [14 out of the total 69 subjects had provided sufficient concentration-time data for PK analysis and estimating the PK parameters]
Measure: Mean (Standard Deviation); unit: hours
Groups:
- Asfotase Alfa: A total of 6 mg/kg/week of asfotase alfa administered by SC injection (2 mg/kg asfotase alfa 3 times per week)
Arm/Group | Asfotase Alfa
Number analyzed (Participants) | 14
hours | 48.1 (0.1)

13. Secondary Outcome: Pharmacokinetic (PK) Properties of Asfotase Alfa (Tmax)
Description: The PK properties (tmax) of asfotase alfa
Time Frame: as for outcome 12
Population: 14 out of the total 69 subjects had provided sufficient concentration-time data for PK analysis and estimating the PK parameters
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Asfotase Alfa
Number analyzed (Participants) | 14
hours | 14.9 (10.4)

14. Secondary Outcome: Pharmacokinetic (PK) Properties of Asfotase Alfa (Cmax)
Description: The PK properties (Cmax) of asfotase alfa
Time Frame: as for outcome 12
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Asfotase Alfa
Number analyzed (Participants) | 14
ng/mL | 1794 (690)

15. Secondary Outcome: Pharmacokinetic (PK) Properties of Asfotase Alfa (AUCt)
Description: The PK properties (AUCt) of asfotase alfa
Time Frame: as for outcome 12
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | Asfotase Alfa
Number analyzed (Participants) | 14
h*ng/mL | 66042 (25758)

ADVERSE EVENTS:
Time Frame: Starting after signing of informed consent through 30 days after the EOS visit, approximately 6 years
Arm/Group | Asfotase Alfa
All-Cause Mortality (participants affected / at risk) | 9/69
Serious Adverse Events (participants affected / at risk) | 50/69
Other Adverse Events (participants affected / at risk) | 68/69
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Asfotase Alfa (N=69)
Pneumonia (Infections and infestations) | 8 (9)
Pneumonia viral (Infections and infestations) | 3 (3)
Device related infection (Infections and infestations) | 2 (5)
Gastroenteritis (Infections and infestations) | 2 (2)
Gastroenteritis rotavirus (Infections and infestations) | 2 (2)
Respiratory syncytial virus infection (Infections and infestations) | 2 (2)
Rhinovirus infection (Infections and infestations) | 2 (3)
Sepsis (Infections and infestations) | 2 (2)
Upper respiratory tract infection (Infections and infestations) | 2 (2)
Viral infection (Infections and infestations) | 2 (2)
Viral upper respiratory tract infection (Infections and infestations) | 2 (2)
Adenoviral upper respiratory infection (Infections and infestations) | 1 (1)
Bacteraemia (Infections and infestations) | 1 (2)
Beta haemolytic streptococcal infection (Infections and infestations) | 1 (1)
Bronchiolitis (Infections and infestations) | 1 (1)
Bronchitis (Infections and infestations) | 1 (1)
Clostridium difficile colitis (Infections and infestations) | 1 (1)
Corona virus infection (Infections and infestations) | 1 (1)
Enterobacter infection (Infections and infestations) | 1 (1)
Gastroenteritis viral (Infections and infestations) | 1 (1)
Influenza (Infections and infestations) | 1 (1)
Lower respiratory tract infection (Infections and infestations) | 1 (1)
Meningitis staphylococcal (Infections and infestations) | 1 (1)
Otitis media (Infections and infestations) | 1 (2)
Parainfluenzae virus infection (Infections and infestations) | 1 (1)
Postoperative wound infection (Infections and infestations) | 1 (1)
Pseudomonas infection (Infections and infestations) | 1 (1)
Respiratory tract infection (Infections and infestations) | 1 (1)
Respiratory tract infection viral (Infections and infestations) | 1 (1)
Serratia infection (Infections and infestations) | 1 (1)
Serratia sepsis (Infections and infestations) | 1 (1)
Staphylococcal infection (Infections and infestations) | 1 (1)
Staphylococcal sepsis (Infections and infestations) | 1 (1)
Stenotrophomonas infection (Infections and infestations) | 1 (1)
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 4 (6)
Apnoea (Respiratory, thoracic and mediastinal disorders) | 3 (5)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 3 (4)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (3)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (8)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Adenoidal hypertrophy (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Collapse of lung (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (5)
Obstructive airways disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 1 (3)
Craniosynostosis (Congenital, familial and genetic disorders) | 13 (13)
Arnold-Chiari malformation (Congenital, familial and genetic disorders) | 3 (5)
Hypophosphatasia (Congenital, familial and genetic disorders) | 1 (1)
Hydrocephalus (Nervous system disorders) | 3 (4)
Intracranial pressure increased (Nervous system disorders) | 3 (3)
Syringomyelia (Nervous system disorders) | 3 (3)
Convulsion (Nervous system disorders) | 2 (2)
Headache (Nervous system disorders) | 2 (2)
Brain oedema (Nervous system disorders) | 1 (1)
Encephalitis (Nervous system disorders) | 1 (1)
Febrile convulsion (Nervous system disorders) | 1 (2)
Haemorrhagic stroke (Nervous system disorders) | 1 (1)
Intracranial hypotension (Nervous system disorders) | 1 (1)
Motor developmental delay (Nervous system disorders) | 1 (1)
Motor dysfunction (Nervous system disorders) | 1 (1)
Neurological symptom (Nervous system disorders) | 1 (1)
Petit mal epilepsy (Nervous system disorders) | 1 (1)
Oxygen saturation decreased (Investigations) | 4 (14)
Aspiration tracheal (Investigations) | 1 (1)
CSF pressure (Investigations) | 1 (1)
Enterovirus test positive (Investigations) | 1 (1)
Hepatic enzyme increased (Investigations) | 1 (1)
Human rhinovirus test positive (Investigations) | 1 (1)
Neurological examination abnormal (Investigations) | 1 (1)
Nuclear magnetic resonance imaging (Investigations) | 1 (1)
Respiratory rate increased (Investigations) | 1 (1)
Respiratory syncytial virus test positive (Investigations) | 1 (1)
Weight decreased (Investigations) | 1 (1)
Pyrexia (General disorders) | 6 (14)
Irritability (General disorders) | 2 (2)
Chills (General disorders) | 1 (1)
Device dislocation (General disorders) | 1 (1)
Injection site erythema (General disorders) | 1 (2)
Oedema (General disorders) | 1 (1)
Femur fracture (Injury, poisoning and procedural complications) | 3 (3)
Feeding tube complication (Injury, poisoning and procedural complications) | 2 (6)
Abdominal wound dehiscence (Injury, poisoning and procedural complications) | 1 (1)
Brain herniation (Injury, poisoning and procedural complications) | 1 (1)
Endotracheal intubation complication (Injury, poisoning and procedural complications) | 1 (3)
Eye injury (Injury, poisoning and procedural complications) | 1 (1)
Humerus fracture (Injury, poisoning and procedural complications) | 1 (1)
Incorrect dose administered (Injury, poisoning and procedural complications) | 1 (1)
Rib fracture (Injury, poisoning and procedural complications) | 1 (1)
Food intolerance (Metabolism and nutrition disorders) | 4 (5)
Failure to thrive (Metabolism and nutrition disorders) | 2 (3)
Feeding disorder (Metabolism and nutrition disorders) | 2 (2)
Hyponatraemia (Metabolism and nutrition disorders) | 2 (2)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Dystrophic calcification (Metabolism and nutrition disorders) | 1 (1)
Fluid overload (Metabolism and nutrition disorders) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1)
Hypernatraemia (Metabolism and nutrition disorders) | 1 (1)
Hyperphosphataemia (Metabolism and nutrition disorders) | 1 (1)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1)
Hypophagia (Metabolism and nutrition disorders) | 1 (2)
Hypervolaemia (Metabolism and nutrition disorders) | 1 (1)
Bradycardia (Cardiac disorders) | 3 (10)
Cardio-respiratory arrest (Cardiac disorders) | 2 (4)
Cardiac arrest (Cardiac disorders) | 3 (4)
Cyanosis (Cardiac disorders) | 2 (3)
Arrhythmia (Cardiac disorders) | 1 (1)
Cardiopulmonary failure (Cardiac disorders) | 1 (1)
Wolff-Parkinson-White syndrome (Cardiac disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 3 (4)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1)
Inguinal hernia (Gastrointestinal disorders) | 1 (1)
Pancreatitis acute (Gastrointestinal disorders) | 1 (1)
Pneumatosis intestinalis (Gastrointestinal disorders) | 1 (1)
Rectal prolapse (Gastrointestinal disorders) | 1 (2)
Osteopenia (Musculoskeletal and connective tissue disorders) | 2 (3)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Joint contracture (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1)
Pathological fracture (Musculoskeletal and connective tissue disorders) | 1 (1)
Cranial operation (Surgical and medical procedures) | 1 (1)
Medical device removal (Surgical and medical procedures) | 1 (1)
Tracheal operation (Surgical and medical procedures) | 1 (1)
Tracheostomy (Surgical and medical procedures) | 1 (1)
Wean from ventilator (Surgical and medical procedures) | 1 (1)
Drug hypersensitivity (Immune system disorders) | 2 (2)
Anaphylactoid reaction (Immune system disorders) | 1 (1)
Conjunctivitis (Eye disorders) | 1 (1)
Optic neuropathy (Eye disorders) | 1 (1)
Coagulopathy (Blood and lymphatic system disorders) | 1 (1)
Hyperparathyroidism tertiary (Endocrine disorders) | 1 (1)
Breath holding (Psychiatric disorders) | 1 (1)
Staring (Psychiatric disorders) | 1 (1)
Renal failure (Renal and urinary disorders) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Asfotase Alfa (N=69)
Nasopharyngitis (Infections and infestations) | 18 (52)
Upper respiratory tract infection (Infections and infestations) | 17 (31)
Gastroenteritis (Infections and infestations) | 16 (20)
Respiratory tract infection (Infections and infestations) | 16 (62)
Ear infection (Infections and infestations) | 13 (18)
Rhinitis (Infections and infestations) | 10 (17)
Bronchitis (Infections and infestations) | 9 (16)
Urinary tract infection (Infections and infestations) | 8 (8)
Influenza (Infections and infestations) | 7 (8)
Pneumonia (Infections and infestations) | 7 (9)
Device related infection (Infections and infestations) | 5 (5)
Hand-foot-and-mouth disease (Infections and infestations) | 5 (5)
Otitis media (Infections and infestations) | 5 (5)
Tonsillitis (Infections and infestations) | 5 (5)
Gastroenteritis viral (Infections and infestations) | 4 (5)
Gastrointestinal infection (Infections and infestations) | 4 (9)
Viral upper respiratory tract infection (Infections and infestations) | 4 (4)
Pyrexia (General disorders) | 47 (131)
Injection site erythema (General disorders) | 33 (223)
Injection site discolouration (General disorders) | 12 (43)
Injection site induration (General disorders) | 11 (44)
Injection site haematoma (General disorders) | 10 (22)
Injection site pain (General disorders) | 8 (22)
Injection site reaction (General disorders) | 8 (13)
Injection site swelling (General disorders) | 7 (21)
Injection site pruritus (General disorders) | 6 (14)
Catheter site erythema (General disorders) | 5 (16)
Injection site papule (General disorders) | 5 (91)
Injection site rash (General disorders) | 5 (5)
Catheter site inflammation (General disorders) | 4 (5)
Device occlusion (General disorders) | 4 (8)
Injection site atrophy (General disorders) | 4 (15)
Irritability (General disorders) | 4 (6)
Tooth loss (Gastrointestinal disorders) | 41 (109)
Vomiting (Gastrointestinal disorders) | 30 (92)
Diarrhoea (Gastrointestinal disorders) | 20 (35)
Constipation (Gastrointestinal disorders) | 16 (37)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 9 (10)
Abdominal pain (Gastrointestinal disorders) | 7 (7)
Dental caries (Gastrointestinal disorders) | 7 (11)
Teething (Gastrointestinal disorders) | 5 (10)
Toothache (Gastrointestinal disorders) | 5 (8)
Contusion (Injury, poisoning and procedural complications) | 10 (21)
Fall (Injury, poisoning and procedural complications) | 7 (9)
Arthropod bite (Injury, poisoning and procedural complications) | 5 (5)
Procedural pain (Injury, poisoning and procedural complications) | 5 (6)
Rib fracture (Injury, poisoning and procedural complications) | 5 (5)
Tooth fracture (Injury, poisoning and procedural complications) | 4 (4)
Cough (Respiratory, thoracic and mediastinal disorders) | 17 (34)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 8 (30)
Use of accessory respiratory muscles (Respiratory, thoracic and mediastinal disorders) | 7 (16)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 6 (12)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 6 (7)
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 6 (7)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 5 (6)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 4 (6)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Tracheomalacia (Respiratory, thoracic and mediastinal disorders) | 4 (5)
Rash (Skin and subcutaneous tissue disorders) | 11 (23)
Dermatitis diaper (Skin and subcutaneous tissue disorders) | 10 (18)
Dry skin (Skin and subcutaneous tissue disorders) | 8 (10)
Eczema (Skin and subcutaneous tissue disorders) | 7 (14)
Erythema (Skin and subcutaneous tissue disorders) | 6 (8)
Excessive granulation tissue (Skin and subcutaneous tissue disorders) | 5 (6)
Granuloma skin (Skin and subcutaneous tissue disorders) | 4 (7)
Heat rash (Skin and subcutaneous tissue disorders) | 4 (5)
Alanine aminotransferase increased (Investigations) | 6 (8)
Aspartate aminotransferase increased (Investigations) | 5 (6)
Oxygen saturation decreased (Investigations) | 5 (54)
Vitamin D decreased (Investigations) | 4 (6)
Hypocalcaemia (Metabolism and nutrition disorders) | 6 (8)
Hypoglycaemia (Metabolism and nutrition disorders) | 6 (6)
Hypokalaemia (Metabolism and nutrition disorders) | 6 (7)
Food intolerance (Metabolism and nutrition disorders) | 4 (5)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 11 (13)
Kyphosis (Musculoskeletal and connective tissue disorders) | 6 (10)
Knee deformity (Musculoskeletal and connective tissue disorders) | 5 (5)
Bone disorder (Musculoskeletal and connective tissue disorders) | 4 (23)
Conjunctivitis (Eye disorders) | 8 (16)
Papilloedema (Eye disorders) | 5 (8)
Headache (Nervous system disorders) | 10 (22)
Cerebral ventricle dilatation (Nervous system disorders) | 4 (6)
Craniosynostosis (Congenital, familial and genetic disorders) | 10 (11)
Congenital bowing of long bones (Congenital, familial and genetic disorders) | 5 (6)
Anaemia (Blood and lymphatic system disorders) | 9 (13)
Lymphadenopathy (Blood and lymphatic system disorders) | 5 (7)
Neutropenia (Blood and lymphatic system disorders) | 4 (4)
Nephrocalcinosis (Renal and urinary disorders) | 5 (5)
Agitation (Psychiatric disorders) | 4 (11)
Cerumen impaction (Ear and labyrinth disorders) | 5 (11)
Tachycardia (Cardiac disorders) | 6 (16)
Bradycardia (Cardiac disorders) | 4 (7)
Hypertension (Vascular disorders) | 4 (4)
Hepatomegaly (Hepatobiliary disorders) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less